## Abbreviated Injury Scale (AIS) Grading and Simple Triage and Rapid Treatment (START) Combined with Film Transferring on Instant Message Improve The Difference of Disaster Triage and Disaster Management

NCT number: nil

date of the document: 20220414

**Objectives:** The AIS and START grading are usually defined in trauma disaster when patients are sent off to emergency room. The AIS is an anatomically-based injury severity scoring system that classifies each injury by body region on a 6 point scale from minor to maximal (currently untreatable) status. The START grading assign the disaster patients to one of the following four categories: grade 0:deceased/expectant (black), grade1: immediate (red), grade 2: delayed (yellow), grade 3:minor (green) **Design and Methods:** The investigators use the recorded exterior photo, radiological film and vital sign data of the injured patients to re-define the AIS and START grading. The results will be compared with the original data documented in our medical records and want to know that the consistency exist between two groups. Excluding patients with incomplete clinical data of treatment.